CLINICAL TRIAL: NCT07324057
Title: The Effects of Preoperative Intranasal Administration of Dexmedetomidine and Esketamine on Negative Postoperative Behavioral Changes in Children With Autism Spectrum Disorder
Acronym: NPOBCs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Fei (Other)
Responsible Party: Sponsor-Investigator, Sun Fei, Attending Physician, Nanjing Children's Hospital
Organization: Nanjing Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202504034-2; 202511028 (Other Grant/Funding Number: Nanjing Municipal Science and Technology Bureau)
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Children;Anesthetic agents;Autism Spectrum Disorder;Electroencephalography;Negative postoperative behavioural changes
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study employed a double-blind design for both investigators and patients. Approximately 30 minutes prior to surgery, the paediatric patient was admitted to the anaesthesia preparation room. An anaesthesia nurse not involved in the study received the randomisation allocation results from the centralised system and prepared the corresponding formulations. The study medication was administered via identical, unlabelled nasal spray pumps, All formulations were diluted to 1 ml and then loaded into sterile, unlabelled nasal spray pumps. These were handed to the study intervention implementer, who remained unaware of the administered drug and withdrew from the study upon completion of the intervention. Subsequently, all investigators remained unaware of the group allocation. Postoperative follow-up was conducted by another independent investigator, and data analysis was performed by a statistical expert not involved in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine Intranasal Spray (D Group) (Experimental): Participants assigned to the Dexmedetomidine Intranasal Spray receive dexmedetomidine at a dose of 2 micrograms per kilogram (maximum 100 micrograms), diluted to 1 milliliter and administered intranasally approximately 30 minutes before anesthesia induction.
  Interventions: Drug: Intranasal dexmedetomidine
- Esketamine Intranasal Spray (L Group) (Experimental): Participants receive esketamine 1 milligram per kilogram (maximum 50 milligrams), diluted to 1 milliliter and administered intranasally approximately 30 minutes before anesthesia induction.
  Interventions: Drug: Intranasal Esketamine
- Saline Control Group (C Group) (Placebo Comparator): Participants receive normal saline 1 milliliter administered intranasally approximately 30 minutes before anesthesia induction.
  Interventions: Drug: saline control

INTERVENTIONS:
Drug: Intranasal dexmedetomidine — Dosage: 2.0 µg/kg (maximum 100 µg) Administration: Intranasal spray, 30 minutes before anesthesia induction Purpose: To provide sedation, reduce preoperative anxiety, and potentially prevent postoperative behavioral issues like agitation and delirium.
  Other Names: · Dexmedetomidine nasal spray · Intranasal dexmedetomidine · Dexmedetomidine intranasal spray · Dexmedetomidine intranasal group (D group)
  Arms: Dexmedetomidine Intranasal Spray (D Group)
Drug: Intranasal Esketamine — Dosage: 1.0 mg/kg (maximum 50 mg) Administration: Intranasal spray, 30 minutes before anesthesia induction Purpose: To provide sedation, reduce anxiety, and minimize postoperative behavioral changes like aggression and agitation.
  Other Names: · Esketamine nasal spray · Intranasal esketamine · Esketamine intranasal spray · Esketamine intranasal group (K group)
  Arms: Esketamine Intranasal Spray (L Group)
Drug: saline control — Dosage: Equal volume of saline (1 ml) Administration: Intranasal spray, 30 minutes before anesthesia induction Purpose: To serve as a placebo control, allowing comparison to the active intervention groups.
  Other Names: Normal saline Physiological saline Intranasal saline Normal saline nasal spray (1 mL) Saline control group (C group)
  Arms: Saline Control Group (C Group)

SUMMARY:
The goal of this clinical trial is to learn whether intranasal sedation given before anesthesia can lower negative postoperative behavioral changes in children with autism spectrum disorder who undergo elective surgery. The study will compare two commonly used sedative medicines with a saline control. It will also examine the safety of these medicines and explore how brain electrical activity during recovery may relate to later behavior changes.

The main questions this study aims to answer are:

* Does intranasal dexmedetomidine given before anesthesia lower negative postoperative behavioral changes seven days after surgery in children with autism spectrum disorder?

  * Does intranasal esketamine given before anesthesia lower negative postoperative behavioral changes seven days after surgery in children with autism spectrum disorder?

    * Are there differences in postoperative agitation, pain, and sedation quality among the three groups? Researchers will compare dexmedetomidine, esketamine, and saline to see whether either medicine works better than saline in reducing postoperative behavior changes.

Participants will:

* Be randomly assigned to receive intranasal dexmedetomidine, intranasal esketamine, or intranasal saline about thirty minutes before anesthesia

  * Undergo their planned surgery with standard general anesthesia care ③ Be assessed for behavior changes at three, seven, and twenty-eight days after surgery ④ Have routine monitoring of recovery, pain, agitation, and safety outcomes during and after surgery

DETAILED DESCRIPTION:
This study is a multicenter, prospective, randomized, double-blind, controlled clinical trial designed to evaluate the effects of preoperative intranasal sedation on negative postoperative behavioral changes (NPOBCs) in children with autism spectrum disorder (ASD) undergoing elective surgery under general anesthesia Children with ASD often experience heightened perioperative anxiety, sensory sensitivity, and difficulty adapting to unfamiliar medical environments. These factors place them at increased risk for NPOBCs, which may include emotional distress, irritability, sleep disturbances, fear-related behaviors, and reduced cooperation with medical care after surgery. Effective and well-tolerated preoperative sedation may help reduce perioperative stress responses and improve postoperative behavioral outcomes. However, high-quality evidence in children with ASD remains limited.

This study will enroll a total of 234 participants across multiple pediatric hospitals. Participants will be randomly assigned in a 1:1:1 ratio to one of three intervention groups: intranasal dexmedetomidine, intranasal esketamine, or intranasal saline as a control. Randomization will be centrally managed using a stratified block design to balance study center, age group, and surgical category. Blinding will be maintained for participants, caregivers, anesthesiologists, outcome assessors, and data analysts to minimize bias.

Study medication will be administered intranasally approximately thirty minutes before anesthesia induction using identical, unlabeled nasal spray devices. All participants will then receive routine general anesthesia and perioperative management according to standard clinical practice at each participating center. The surgical procedure and anesthetic technique will not be altered by study participation.

The primary objective of the study is to compare the incidence of NPOBCs seven days after surgery among the three groups. Behavioral outcomes will be assessed using validated caregiver-reported questionnaires appropriate for children with ASD. Secondary objectives include evaluating behavioral changes at three and twenty-eight days after surgery, emergence agitation during recovery, postoperative pain, quality of preoperative sedation, and overall safety.

In addition to clinical and behavioral assessments, electroencephalographic (EEG) data will be collected during the emergence period from anesthesia. These data will be analyzed to explore potential associations between neurophysiological patterns and subsequent behavioral outcomes. This exploratory component aims to support the development of predictive models for postoperative behavioral risk in children with ASD.

Participant safety is a key priority. All adverse events will be systematically recorded and reviewed in accordance with Good Clinical Practice guidelines. Serious adverse events will be reported promptly and reviewed by an independent data and safety monitoring process. Ongoing safety oversight will include regular review of adverse event rates across study centers.

The study is expected to provide clinically relevant evidence on whether intranasal dexmedetomidine or intranasal esketamine administered before anesthesia can reduce postoperative behavioral disturbances in children with ASD. Findings from this trial may help inform future perioperative management strategies and support more individualized, evidence-based care for this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-12 years ASA physical status I-III Diagnosed with Autism Spectrum Disorder (ASD) by a psychiatrist Scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* Cardiac, thoracic/pulmonary, or neurosurgery Congenital disease or severe hepatic/renal dysfunction Allergy to study drugs Neuromuscular disease, cerebral palsy, or epilepsy Other psychiatric or neurologic disorders BMI ≥30 kg/m² Severe upper respiratory tract infection preoperatively Sedatives or analgesics used within 48 hours preoperatively Major life stressor within 1 month pre-op (e.g., family/school change, parental divorce or death) Parent/guardian refuses participation

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 234 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of negative postoperative behavioral changes (NPOBCs) at postoperative day 7, assessed using the Post Hospitalization Behavior Questionnaire for Autism Spectrum Disorder (PHBQ-AS). | Postoperative day 7
  Incidence of negative postoperative behavioral changes (NPOBCs) at postoperative day 7, assessed using the Post Hospitalization Behavior Questionnaire for Ambulatory Surgery (PHBQ-AS). NPOBCs refer to new or worsened maladaptive behaviors after anesthesia/surgery (e.g., sleep disturbance, changes in eating behavior, emotional dysregulation such as irritability/anxiety, and medical-related fears). The day-7 PHBQ-AS assessment will be collected during postoperative follow-up performed by an independent researcher who is blinded to group allocation.

SECONDARY OUTCOMES:
Incidence of negative postoperative behavioral changes (NPOBCs) at postoperative day 1 and postoperative day 30, assessed using the Post Hospitalization Behavior Questionnaire for Autism Spectrum Disorder (PHBQ-AS). | Postoperative day 3 and postoperative day 28
  Incidence of negative postoperative behavioral changes (NPOBCs) at postoperative day 3 and postoperative day 28, assessed using the Post Hospitalization Behavior Questionnaire for Autism Spectrum Disorder (PHBQ-AS) during postoperative follow-up. NPOBCs are defined as new or worsened maladaptive behaviors after anesthesia/surgery, which may include changes such as sleep disturbance, altered eating patterns, emotional dysregulation (e.g., irritability/anxiety), medical-related fears, and reduced treatment cooperation. Follow-up assessments are performed by an independent researcher blinded to group allocation.

OTHER OUTCOMES:
Additional protocol-defined outcome measures collected and analyzed as planned, but not labeled primary or secondary (e.g., exploratory/tertiary); exclude post-hoc measures. | From 30 minutes after study drug administration through surgery, emergence/awakening, and the postoperative hospital stay (until discharge).
  This trial's other pre-specified outcomes include: sedation 30 minutes after study drug administration measured with MOAA/S; pain after awakening measured with FLACC; emergence delirium/agitation after awakening measured with PAED; intraoperative and emergence EEG features; perioperative adverse events (e.g., nausea/vomiting, allergy); awakening time and postoperative length of stay; and parent satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
At this time, there are no plans to share individual participant data (IPD) from this study. The decision may be revisited in the future based on data confidentiality, privacy concerns, and any relevant regulatory requirements.

DOCUMENTS (2):
  • Study Protocol (2025-05-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT07324057/Prot_000.pdf
  • Informed Consent Form (2025-05-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT07324057/ICF_001.pdf